CLINICAL TRIAL: NCT01681095
Title: Custodiol-HTK Solution as a Cardioplegic Agent- A Prospective Non-Inferiority Randomized Clinical Trial
Brief Title: Custodiol-HTK (Histidine-tryptophan-ketoglutarate) Solution as a Cardioplegic Agent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marc Sakwa, MD (Other)
Collaborators: Essential Pharmaceuticals, LLC (Other)
Responsible Party: Sponsor-Investigator, Marc Sakwa, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-125
Record Dates: First submitted 2012-08-10; First posted 2012-09-07 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2017-01

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Valvular Heart Disease
Keywords: Physiological Effects of Drugs; Cardiovascular Agents; Therapeutic Uses; Pharmacologic Actions; Mannitol; Cardiac Surgery; Cardioplegic Solutions; HTK solution; Myocardial protection; Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Heart Valve Diseases | interventions — Bretschneider cardioplegic solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardioplegia: Custodiol HTK Solution (Experimental): Custodiol HTK (histidine-tryptophan-ketoglutarate) cardioplegia: One liter of HTK solution (Custodiol; Koehler Chemi, Alsbach-Haenlien, Germany) contains the following components: 15 mmol/L sodium chloride, 9 mmol/L potassium chloride, 4 mmol/L magnesium chloride, 18 mmol/L histidine hydrochloride, 180 mmol/L histidine, 2 mmol/L tryptophan, 30 mmol/L mannitol, 0.015 mmol/L calcium chloride, 1 mmol/L potassium hydrogen 2-ketoglutarate, osmolarity 310 mOsm/kg, pH 7.02-7.20.
  Custodiol-HTK was delivered to establish and maintain cardiac arrest. After cross-clamping of the aorta approximately 1-2 L of Custodiol-HTK was infused into the ascending aorta over 6-8 minutes. Additional doses of 100-200 ml were administered as needed. Custodiol-HTK was delivered at a temperature of 4°C - 10°C.
  Interventions: Drug: Custodiol HTK
- Cold Blood Cardioplegia (Active Comparator): Cold Blood Cardioplegia: One liter of cold blood cardioplegic solution, mixed at a ratio of 4:1 per Beaumont standard of care (blood /cardioplegic solution), contains the following in a 500 cc bag of D5W (dextrose 5% in water): 50meq/L potassium chloride, 37.5 meq/L sodium bicarbonate and 7.5 meq/L magnesium sulfate.
  After cross-clamping the aorta, at least 1000 mL of a 4:1 mixture of cold blood: cold crystalloid was administered at a pressure of 300 mmHg or less via a twin roller pump. Every 20 minutes an additional > 200 mL was administered as needed. The cardioplegic solution was delivered at a temperature of 4°C - 8°C.
  Interventions: Drug: Cold Blood Cardioplegia

INTERVENTIONS:
Drug: Custodiol HTK — After cross-clamping of the aorta approximately 1-2 L of Custodiol-HTK was infused into the ascending aorta over 6-8 minutes. Additional doses of 100-200 ml were administered as needed. The cardioplegic solution was delivered at a temperature of 4°C - 10°C.
  Other Names: Histidine-tryptophan-ketoglutarate cardioplegia solution
  Arms: Cardioplegia: Custodiol HTK Solution
Drug: Cold Blood Cardioplegia — After cross-clamping the aorta, at least 1000 mL of a 4:1 mixture of cold blood: cold crystalloid was administered at a pressure of 300 mmHg or less via a twin roller pump. Every 20 minutes an additional > 200 mL was administered in an antegrade/retrograde fashion throughout the remainder of the case. The cardioplegic solution was delivered at a temperature of 4°C - 8°C.
  Arms: Cold Blood Cardioplegia

SUMMARY:
The purpose of the study is to demonstrate that Custodiol-HTK is not inferior to cold cardioplegic solution in patients undergoing cardiovascular surgery requiring cardioplegic arrest.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate that Custodiol is not inferior to cold cardioplegic solution for myocardial protection by comparing standard cold blood cardioplegia to Custodiol solution with respect to myocardial injury as measured by Creatine phosphokinase MB isoenzyme (CK-MB),troponin-I at 7 hours post surgery and changes in ejection fraction by trans-thoracic echocardiogram (TTE)or trans-esophageal echocardiogram (TEE) at 24 hours post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled cardiac surgery requiring cardioplegic arrest with expected cross clamp time>45 minutes
* Patients age 18 and older

Exclusion Criteria:

* Pregnant women*
* Urgent or emergent cases
* Repeat cardiovascular surgical procedures
* Patients on dialysis
* Any known allergies to components of either cardioplegia solution *All women of child bearing potential must have a negative serum or urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sakwa, M.D., Principal Investigator — Beaumont Health
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braathen B, Jeppsson A, Schersten H, Hagen OM, Vengen O, Rexius H, Lepore V, Tonnessen T. One single dose of histidine-tryptophan-ketoglutarate solution gives equally good myocardial protection in elective mitral valve surgery as repetitive cold blood cardioplegia: a prospective randomized study. J Thorac Cardiovasc Surg. 2011 Apr;141(4):995-1001. doi: 10.1016/j.jtcvs.2010.07.011. Epub 2010 Aug 30. PMID 20800244
- [Background] Careaga G, Salazar D, Tellez S, Sanchez O, Borrayo G, Arguero R. Clinical impact of histidine-ketoglutarate-tryptophan (HTK) cardioplegic solution on the perioperative period in open heart surgery patients. Arch Med Res. 2001 Jul-Aug;32(4):296-9. doi: 10.1016/s0188-4409(01)00296-x. PMID 11440787
- [Background] Hachida M, Ookado A, Nonoyama M, Koyanagi H. Effect of HTK solution for myocardial preservation. J Cardiovasc Surg (Torino). 1996 Jun;37(3):269-74. PMID 8698763
- [Background] Yang Q, He GW. Effect of cardioplegic and organ preservation solutions and their components on coronary endothelium-derived relaxing factors. Ann Thorac Surg. 2005 Aug;80(2):757-67. doi: 10.1016/j.athoracsur.2004.10.003. PMID 16039259
- [Background] Beyersdorf F, Krause E, Sarai K, Sieber B, Deutschlander N, Zimmer G, Mainka L, Probst S, Zegelman M, Schneider W, et al. Clinical evaluation of hypothermic ventricular fibrillation, multi-dose blood cardioplegia, and single-dose Bretschneider cardioplegia in coronary surgery. Thorac Cardiovasc Surg. 1990 Feb;38(1):20-9. doi: 10.1055/s-2007-1013985. PMID 2106735
- [Background] Savini C, Camurri N, Castelli A, Dell'Amore A, Pacini D, Suarez SM, Grillone G, Di Bartolomeo R. Myocardial protection using HTK solution in minimally invasive mitral valve surgery. Heart Surg Forum. 2005;8(1):E25-7. doi: 10.1532/HSF98.20041145. PMID 15769709
- [Background] Braathen B, Tonnessen T. Cold blood cardioplegia reduces the increase in cardiac enzyme levels compared with cold crystalloid cardioplegia in patients undergoing aortic valve replacement for isolated aortic stenosis. J Thorac Cardiovasc Surg. 2010 Apr;139(4):874-80. doi: 10.1016/j.jtcvs.2009.05.036. Epub 2009 Jul 26. PMID 19660338
- [Background] Hendrikx M, Jiang H, Gutermann H, Toelsie J, Renard D, Briers A, Pauwels JL, Mees U. Release of cardiac troponin I in antegrade crystalloid versus cold blood cardioplegia. J Thorac Cardiovasc Surg. 1999 Sep;118(3):452-9. doi: 10.1016/s0022-5223(99)70182-0. PMID 10469959
- [Background] Aarsaether E, Stenberg TA, Jakobsen O, Busund R. Mechanoenergetic function and troponin T release following cardioplegic arrest induced by St Thomas' and histidine-tryptophan-ketoglutarate cardioplegia--an experimental comparative study in pigs. Interact Cardiovasc Thorac Surg. 2009 Oct;9(4):635-9. doi: 10.1510/icvts.2009.208231. Epub 2009 Jul 23. PMID 19628529
- [Background] Gallandat Huet RC, Karliczek GF, van der Heide JN, Brenken U, Mooi B, van der Broeke JJ, Jenkins I, de Geus AF. Clinical effect of Bretschneider-HTK and St. Thomas cardioplegia on hemodynamic performance after bypass measured using an automatic datalogging database system. Thorac Cardiovasc Surg. 1988 Jun;36(3):151-6. doi: 10.1055/s-2007-1020064. PMID 3145585
- [Background] Arslan A, Sezgin A, Gultekin B, Ozkan S, Akay T, Uguz E, Tasdelen A, Aslamaci S. Low-dose histidine-tryptophan-ketoglutarate solution for myocardial protection. Transplant Proc. 2005 Sep;37(7):3219-22. doi: 10.1016/j.transproceed.2005.08.020. PMID 16213352
- [Background] Fannelop T, Dahle GO, Salminen PR, Moen CA, Matre K, Mongstad A, Eliassen F, Segadal L, Grong K. Multidose cold oxygenated blood is superior to a single dose of Bretschneider HTK-cardioplegia in the pig. Ann Thorac Surg. 2009 Apr;87(4):1205-13. doi: 10.1016/j.athoracsur.2009.01.041. PMID 19324152
- [Background] Schaper J, Scheld HH, Schmidt U, Hehrlein F. Ultrastructural study comparing the efficacy of five different methods of intraoperative myocardial protection in the human heart. J Thorac Cardiovasc Surg. 1986 Jul;92(1):47-55. PMID 3088335
- [Background] Athanasuleas C., Buckberg G. Myocardial protection and cardioplegia. Cardiopulmonary Bypass. New York: CambridgeUniversity Press; 2009: p. 82.
- [Background] Bical OM, Fromes Y, Paumier D, Gaillard D, Foiret JC, Trivin F. Does warm antegrade intermittent blood cardioplegia really protect the heart during coronary surgery? Cardiovasc Surg. 2001 Apr;9(2):188-93. doi: 10.1016/s0967-2109(00)00087-9. PMID 11250190
- [Background] Allen BS, Winkelmann JW, Hanafy H, Hartz RS, Bolling KS, Ham J, Feinstein S. Retrograde cardioplegia does not adequately perfuse the right ventricle. J Thorac Cardiovasc Surg. 1995 Jun;109(6):1116-24; discussion 1124-6. doi: 10.1016/S0022-5223(95)70195-8. PMID 7776676
- [Background] Sakata J, Morishita K, Ito T, Koshino T, Kazui T, Abe T. Comparison of clinical outcome between histidine-triptophan-ketoglutalate solution and cold blood cardioplegic solution in mitral valve replacement. J Card Surg. 1998 Jan;13(1):43-7. doi: 10.1111/j.1540-8191.1998.tb01053.x. PMID 9892485
- [Background] Lee D. H., Park N. H., Keum D. Y., Choi S. Y., Lee K. S., Yoo Y. S. Comparison of Myocardial Protective Effect between the Cold Blood Cardioplegia and Histidine-Tryptophan-Ketoglutarate Solution.Korean J Thorac Cardiovasc Surg. 2004;37(9):739-41.
- [Background] Kim S. , Lee Y. S. , Woo J. S. , Sung S. C. , Choi P. J. , Cho G. J., Bang J. H., Roh M. S. Histidine-tryptophan-ketoglutarate Versus Blood Cardioplegic Solutions: A Prospective, Myocardial Ultrastructural Study.Korean J Thorac Cardiovasc Surg. 2007;40(1):8-16.
- [Background] Choi Y. S., Bang S. O. , Chang B. C. , Lee S. , Park C. H. , Kwak Y. L. A Comparison of the Effects of Histidine-tryptophan-ketoglutarate Solution versus Cold Blood Cardioplegic Solution on Myocardial Protection in Mitral Valve Surgery.Korean J Thorac Cardiovasc Surg. 2007;40(6):399-406
- [Background] Asano H, Kyo S, Ogiwara M, Tsunemoto M, Yokote Y, Omoto R, Koike K, Kobayashi T, Kobayashi J, Taketazu M. [Single-dose and high-volume Bretschneider cardioplegic solution for congenital heart surgery]. Kyobu Geka. 1999 Jan;52(1):82-6. Japanese. PMID 10024809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Cold Blood Cardioplegia: 55 participants were randomized to Standard cold blood cardioplegia. Cold Blood Cardioplegia: One liter of cold blood cardioplegic solution, mixed at a ratio of 4:1 per Beaumont standard of care (blood /cardioplegic solution), contains the following in a 500 cc bag of D5W (dextrose 5% in water): 50meq/L potassium chloride, 37.5 meq/L sodium bicarbonate and 7.5 meq/L magnesium sulfate.
  After cross-clamping the aorta, at least 1000 mL of a 4:1 mixture of cold blood: cold crystalloid was administered at a pressure of 300 mmHg or less via a twin roller pump. Every 20 minutes an additional > 200 mL was administered as needed. The cardioplegic solution was delivered at a temperature of 4°C - 8°C.
- Custiodiol HTK: 55 participants were randomized to Custodiol HTK. Custodiol HTK (histidine-tryptophan-ketoglutarate) cardioplegia: One liter of HTK solution (Custodiol; Koehler Chemi, Alsbach-Haenlien, Germany) contains the following components: 15 mmol/L sodium chloride, 9 mmol/L potassium chloride, 4 mmol/L magnesium chloride, 18 mmol/L histidine hydrochloride, 180 mmol/L histidine, 2 mmol/L tryptophan, 30 mmol/L mannitol, 0.015 mmol/L calcium chloride, 1 mmol/L potassium hydrogen 2-ketoglutarate, osmolarity 310 mOsm/kg, pH 7.02-7.20.
  Custodiol-HTK was delivered to establish and maintain cardiac arrest. After cross-clamping of the aorta approximately 1-2 L of Custodiol-HTK was infused into the ascending aorta over 6-8 minutes. Additional doses of 100-200 ml were administered as needed. Custodiol-HTK was delivered at a temperature of 4°C - 10°C.
- Total: Total of all reporting groups
Arm/Group | Standard Cold Blood Cardioplegia | Custiodiol HTK | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (11) | 63 (13) | 66 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 35 | 29 | 64
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change in Creatine Phosphokinase-MB Isoenzyme (CK-MB)
Description: Creatine phosphokinase MB isoenzyme (CK-MB) difference from baseline 7 hours post surgery
Time Frame: Baseline and 7 hours post surgery
Population: Patients for which both baseline and 7 hours post surgery values were available
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 40 | 38
ng/mL | 18.8 [12.5 to 24] | 22.2 [15 to 51]

2. Primary Outcome: Change in Troponin I
Description: Troponin I values, difference from baseline 7 hours post surgery
Time Frame: Baseline and 7 hours post surgery
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
ng/mL | 9.65 [5.47 to 16.00] | 10.15 [6.04 to 19.97]

3. Primary Outcome: Changes in Left Ventricular (LV) Ejection Fraction (EF) by Transthoracic Echocardiogram (TTE)
Description: LV ejection fraction by TTE, difference from baseline at 24 hours post surgery
Time Frame: Baseline and 24 hours post surgery
Population: patients for whom both preoperative and 24 hour LV ejection fractions were obtained
Measure: Mean (Standard Deviation); unit: % LV volume
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 51 | 51
% LV volume | -0.06 (11) | 1.9 (10)

4. Secondary Outcome: Cardiac Dysrhythmias
Description: Number of participants with new or worsening of cardiac dysrhythmias
Time Frame: up to 36 hrs post surgery
Measure: Number; unit: participants
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
participants | 24 | 30

5. Secondary Outcome: All Cause Mortality
Description: Number of participants with all-cause mortality AS reported in the Society of Thoracic Surgeons (STS) database after 30 days postoperative
Time Frame: 30 days post procedure
Measure: Number; unit: participants
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
participants | 0 | 0

6. Secondary Outcome: Cardiovascular Mortality
Description: Number of participants with cardiovascular-related mortality AS reported in the Society of Thoracic Surgeons (STS) database after 30 days postoperative
Time Frame: 30 days post procedure
Measure: Number; unit: participants
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
participants | 0 | 0

7. Secondary Outcome: Time on Mechanically Assisted Ventilation
Description: time in hours from intubation to extubation, with intervening transport to the cardiac critical care unit.
Time Frame: up to 36 hours post procedure
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
hours | 10.5 [9.1 to 13.9] | 11.4 [3.9 to 527]

8. Secondary Outcome: Duration of Vasopressor / Inotropic Agent
Description: Total time in minutes on any vasopressor or inotropic agent, including norepinephrine, epinephrine, vasopressin, milrinone, dobutamine, dopamine and/or neo-synephrine
Time Frame: up to 36 hours post procedure
Population: Patients not receiving any vasopressors are excluded from this analysis
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 47 | 43
minutes | 340 [115 to 636] | 582 [154 to 1182]

9. Secondary Outcome: Postoperative Inotropic Infusion >20 Minutes
Description: Number of patients receiving vasopressor or inotropic infusion for greater than 20 minutes in the operating room, including norepinephrine, epinephrine, vasopressin, milrinone, dobutamine, dopamine and/or neo-synephrine.
Time Frame: during operative procedure
Measure: Number; unit: participants
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
participants | 47 | 43

10. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: Duration of stay in ICU, from ICU admission to ICU discharge
Time Frame: up to 100 days after admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
days | 3 [2 to 5] | 3 [2 to 5]

11. Secondary Outcome: Myocardial Infarction
Description: Number or participants fulfilling at least two of the following 3 criteria: (1) CK-MB of 100 ug/L or more and/or troponin-I of 3.0 ug/L or more, (2) appearance of new postoperative Q waves on the EKG of more than 0.03 seconds, and (3) a new hypokinetic or akinetic area in the left or right ventricle by echocardiography.
Time Frame: up to 36 hours post procedure
Measure: Number; unit: participants
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 55 | 55
participants | 0 | 0

12. Secondary Outcome: Biochemical Marker - Creatine Kinase MB Isoenzyme (CK-MB)
Description: CK-MB measured pre-operatively
Time Frame: pre-operative
Population: Only patients for whom preoperative CK-MB levels were available were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 38 | 40
ng/mL | 1.9 (1.2) | 2.6 (2.0)

13. Secondary Outcome: Biochemical Marker - Creatine Kinase MB Isoenzyme (CK-MB)
Description: CK-MB measured 24 hours post-operatively
Time Frame: 24 hours post procedure
Population: Only patients for whom 24 hour CK-MB values were available were analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 53 | 54
ng/mL | 20 (14) | 24 (25)

14. Secondary Outcome: Biochemical Marker - Creatine Kinase MB Isoenzyme (CK-MB)
Description: CK-MB measured 48 hours post-operatively
Time Frame: 48 hours post procedure
Population: Only patients for whom 48 hour CK-MB values are available are included in analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 49 | 52
ng/mL | 6.0 (5.1) | 7.8 (7.0)

15. Secondary Outcome: Cardiac Marker - Troponin-I
Description: Troponin-I measured pre-operatively
Time Frame: pre-operatively
Population: Only patients for whom preoperative Troponin-I values were available were included in analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 52 | 54
ng/mL | .03 (.01) | .03 (.01)

16. Secondary Outcome: Cardiac Marker - Troponin-I
Description: Troponin-I measured 24 hours post-operative
Time Frame: 24 hours post procedure
Population: Only patients for whom 24-hour Troponin-I values were available were included in analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 54 | 54
ng/mL | 5.7 (5.4) | 7.8 (8.1)

17. Secondary Outcome: Cardiac Marker - Troponin-I
Description: Troponin-I measured 48 hours post-operative
Time Frame: 48 hours post procedure
Population: Only patients for whom 48-hour Troponin-I values were available were included in analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Number analyzed (Participants) | 49 | 52
ng/mL | 3.0 (3.3) | 4.8 (6.5)

ADVERSE EVENTS:
Time Frame: AEs were evaluated from time of consent to 4 days after surgery.
Description: An assessment of medical records and case report forms were examined for AEs or SAEs. Reports were reviewed by the PI for accuracy and relation to study intervention.
Arm/Group | Cardioplegia: Custodiol HTK Solution | Cold Blood Cardioplegia
Serious Adverse Events (participants affected / at risk) | 3/55 | 9/55
Other Adverse Events (participants affected / at risk) | 25/55 | 34/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioplegia: Custodiol HTK Solution (N=55) | Cold Blood Cardioplegia (N=55)
Profuse bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Approximately 2 hours post-op the subject returned to the OR for re-exploration, finding right ventricular tear. This event was unexpected, and no action was taken with repect to the study drug.
Acute Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Dx 2 days post-op requiring reintubation on 12/19/2012, resolving 1/17/2013, considered an SAE due to prolonged hospitalization, impairment of body structure or body function (Trach on 12/23/2012), unexpected, possibly related to underlying disease.
Acute chest pain, shortness of breath (Cardiac disorders) | 0 (0) | 1 (1) — ER via EMS, L sided chest pain and SOB. Cardiac eval performed. ECG, chest x-ray and labs normal. Admitted for evaluation; the condition resolved. SAE due to hospitalization; unexpected, not related to drug, probably related to underlying disease.
Atrial Fib with rapid ventricular response (Cardiac disorders) | 0 (0) | 1 (1) — PO day 8, EC visit for weakness, ECG demonstrates A-fib w/RVR. Remained in observation, sx resolving within24 hours.SAE due to hospitalization, possibly r/t cardioplegia and possibly underlying disease, unexpected event
SOB, peripheral edema, mouth pain 16 days post-op (Immune system disorders) | 0 (0) | 1 (1) — Subject to ER via EMS. Con-med: Levaquin for pneumonia. Con-med change after evaluation. Resolving after 14days. Possibly r/t study compound, and an unexpected event.
Mediastinal bleed (Surgical and medical procedures) | 0 (0) | 1 (1) — Mediastinal bleed repaired day of surgery and considered resolved. Not related to treatment, possible related to underlying disease and unexpected.
Hospitalization (Infections and infestations) | 0 (0) | 1 (1) — Direct admit from follow-up appt. Fatigue, R groin incision weeping, Atrial flutter w/RVR. Con-med change for incision. Cardioversion. SAE for hospitalization. Resolved and doubtful related to study compound, possible underlying disease.
CVA (Vascular disorders) | 1 (1) | 0 (0) — 1 day post-op, head CT for stroke like sx showing acute cerebral infarct. Con-med changes for L Carotid 30-50% narrowing. Not related to study compound, not related to underlying disease, unexpected. Resolved with sequelae within 9 days.
Community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — ER presentation with hospital admission. Chest x-ray confirming dx. Con-med change. SAE due to hospitalization, not related to study compound, possibly related to underlying disease, unexpected event
Femoral occlusion (Vascular disorders) | 0 (0) | 1 (1) — c/o leg pain, decreased peripheral pulse. 8 days PO performed femoral endarterectomy. Not related to study compound, not related to underlying disease and an unexpected event
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Requiring vent support due to not able to extubate. SAE d/t prolonged hospitalization, not related to study compound, related to underlying disease, an unexpected event.
Emergent Coronary Bypass (Cardiac disorders) | 0 (0) | 1 (1) — Hypoxia, hypotension following MVR. Treated 2 vessels via full sternotomy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cardioplegia: Custodiol HTK Solution (N=55) | Cold Blood Cardioplegia (N=55)
A-Fib or fA-Flutter (Cardiac disorders) | 14 (14) | 21 (21)
Trombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Heart Block (complete, 1st AV, 2 AV, 3 AV) (Cardiac disorders) | 6 (6) | 8 (8)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Bleeding (any) (Surgical and medical procedures) | 5 (5) | 3 (3)
Acute blood loss anemina/any anemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Junctional Rhythm (Cardiac disorders) | 5 (5) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Acute Kidney Failure/Renal Failure (Renal and urinary disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Adverse events (not serious adverse events) are listed only for events occurring with greater than 5% frequency in at least one of the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No